CLINICAL TRIAL: NCT05313958
Title: Treateament of Newly Diagnosed Acute Monocytic Leukemia in Children： A Prospective Multicenter Study in South China
Brief Title: Treateament of Newly Diagnosed Acute Monocytic Leukemia in Children
Acronym: SCCLG-M5
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Maternal and Child Health Hospital of Foshan (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Second Xiangya Hospital of Central South University (Other); Jiangxi Province Children's Hospital (Other); Southern Medical University, China (Other); The First Affiliated Hospital of Nanchang University (Other); Guangzhou First People's Hospital (Other); First Affiliated Hospital of Shantou University Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-052; 2021A1515011809 (Other Grant/Funding Number: Province natural science fund of Guangdong)
Record Dates: First submitted 2021-12-26; First posted 2022-04-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Leukemia, Monocytic, Acute; Pediatric AML
Keywords: Acute monocytic leukemia; pediatric; Cladribine; sorafenib
MeSH Terms: conditions — Leukemia, Monocytic, Acute | interventions — Cladribine; Granulocyte Colony-Stimulating Factor; Cytarabine; Idarubicin; Mitoxantrone; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): The patients in this arm will receive SCCLG-M5 2022 regimen for newly dignosed acute monocytic leukemia (M5) ,including two courses of CLAG(cladribine, darubicin and cytarabine) in the induction period and followed by three courses(HA1M, HA2E, HA3) in consolidation therapy prescribed as the NOPHO-AML 2004 protocol.
  The targeted drugs sorafenib 200mg/m2/day orally is used for FLT3 positive acute monocytic leukemia until molecular biology remission for 2 years.
  Interventions: Drug: Cladribine; Drug: G-CSF; Drug: Cytarabine; Drug: Idarubicin; Drug: Mitoxantrone; Drug: Sorafenib

INTERVENTIONS:
Drug: Cladribine — 5mg/㎡/day d1-5 in 2 hours, before the use of Cytarabine
  Other Names: cladribine injection
Drug: G-CSF — 5ug/kg/day d0-5,if Peripheral blood leukocytes<20,000/ul
  Other Names: granulocyte
Drug: Cytarabine — 2g/㎡/day d1-5 in 4 hours, after the use of Cladribine
  Other Names: Ara-C
Drug: Idarubicin — Idarubicin 10mg/m2/day or mitoxantrone 10mg/m2/day on day 1-3 in the induction therapy II
  Other Names: Idamycin; IDA
Drug: Mitoxantrone — Idarubicin 10mg/m2/day or mitoxantrone 10mg/m2/day on day 1-3 in the induction therapy II
  Other Names: MIT
Drug: Sorafenib — 200mg/m2/day was taken orally until molecular biology remission for 2 years
  Other Names: sorafinib; Nexavar; sorafenib tosylate

SUMMARY:
This is a multicenter, single arm, prospective, intervention trial. Since cladribine can enhance the biological activity and self-protection of cytarabine, giving cladribine and cytarabine together may kill more cancer cells. 10 centers from South China Childhood Leukaemia Collaborative Group carry out the SCCLG-M5-2022 regimen including two courses of CLAG(cladribine, darubicin and cytarabine) in the induction period for the treatment of newly dignosed acute monocytic leukemia (M5). The targeted drugs sorafenib is used for FLT3 positive acute monocytic leukemia to inhibit the serine / threonine kinase activity of FLT3.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

1.To study the 3 year-overall survival of newly diagnosed monocytic leukemia treated with Cladribine and cytarabine in children.

SECONDARY OBJECTIVES

1. To describe the complete response rate following CLAG (cladribine, cytarabine and granulocyte stimulating factor) in newly diagnosed monocytic leukemia in children for intensive induction therapy.
2. To evaluate the 3-year progression-free survival in response to CLAG in children.
3. To assess the toxicity of CLAG including cumulative infection incidence, cumulative adverse effects and chemotherapy-related mortality (TRD).
4. To study the progression-free survival and overall survival (1 year, 2 year and 3 year) of newly diagnosed monocytic leukemia with positive FLT3 treated with CLAG in children and the side effects of sorafenib.

OUTLINE:

1. The induction phase includes two parts including induction therapy I(CLAG) and induction therpay II(CLAG+I/M).
2. The diagnosis and classified criteria is according to the 2016 WHO classification criteria for hematopoietic and lymphoid tissue tumors, and the consolidation therapy consists the therapeutic phases as the NOPHO-AML 2004 protocol prescribed.

   INDUCTION THERAPY I: Patients receive cladribine intravenously (IV) at a dose of 5mg/m2/day combined with cytarabine 2g/m2/day on day 1-5 and granulocyte stimulating factor 5ug/kg/day on day 0-6. When blood count recover(WBC>2.0×109/L， ANC1.0×109/L、PLT≥50×109/L) , Patients achieving a morphological leukemia free state (< 5% blasts) or MRD< 1% receive a second course treatment as above.

   INDUCTION THERPAY II: Patients receive cladribine intravenously (IV) at a dose of 5mg/m2/day combined with cytarabine 2g/m2/day on day 1-5, mitoxantrone/idarubicin 10mg/m2/day on day 1-3 and granulocyte stimulating factor 5ug/kg/day on day 0-6. Patients achieving blast count≥5% or MRD ≥1% proceed to induction II therpy.
3. For FLT3 positive acute monocytic leukemia children, sorafenib 200mg/m2/day was taken orally until molecular biology remission for 2 years.
4. After two courses of indution phase, patients with incomplete response（MRD≥0.1%）are recommended into hematopoietic stem cell transplantation.
5. After two courses of indution phase, patients with persisting positive adverse prognosis cytogenetic abnormalities are recommended into hematopoietic stem cell transplantation.

Patients must meet one of the following risk criteria:

Standard-risk (SR) group meeting all of the following criteria:

Initial WBC < 10,000/μL

M1 (<5%) blasts or MRD<1% in bone marrow after the first course of induction therapy

M1 (<5%) blasts or MRD<0.1% in bone marrow after two courses of induction therapy

Cytogenetic abnormalities with good prognosis

Intermediate-risk (IR) group meeting the following criteria:

Lack of low-risk and high-risk conditions

High-risk (HR) group meeting ≥ 1 of the following criteria:

M2/M3(≥5%) blasts or MRD>5% in bone marrow after the first course of induction therapy

MRD≥0.1% in bone marrow after two course of induction therapy

Cytogenetic abnormalities with poor prognosis

ELIGIBILITY:
Inclusion Criteria:

0-14 years old

Cytologically proven acute monocytic leukemia (M5) with other treatment

Exclusion Criteria:

Secondary to immunodeficiency or MDS

Second tumor

Dowm's syndrome

Evolution of chronic myelogenous leukemia to blast crisis

Death or quit treatment in seven days at the begining of induction therapy

Treatment with other effective chemotherapy drugs for AML, excluding the low dose chemotherapy for the purpose of reducing leukocytes in hyperleukocytic leukemia

Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled heart, brain, liver and kidney failure etc.)

Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 3 years
  TOS was defined as time from diagnostic date through the date of death due to any reasons. For all other participants, the last follow-up available was taken as the last control. If the participant had not completed the study, the date of the last visit available was considered.

SECONDARY OUTCOMES:
Induced remission rate (CR) | 3 years
  According to the time point specified in the treatment plan (22 days after the end of induction I, 29-43 days after the end of induction II and before each consolidation scheme) bone marrow puncture and lumbar puncture were performed. The follow-up contents included the detection of the count of primitive / immature lymphocytes and flow MRD. If there was a positive gene at the onset, the quantitative monitoring of the gene should be performed as MRD data at the same time. If the gene cannot be analyzed quantitatively, PCR qualitative analysis should still be performed as the monitoring basis
Safety,including cumulative infection incidence, adverse reaction and chemotherapy-related mortality (TRD) | 3 years
  During treatment, closely monitor relevant laboratory tests, register adverse reaction records, and report the records according to the requirements of CRF form.
Event-free survival (EFS) | 3 years
  EFS was estimated from date of diagnosis until date of one of the following events: relapse, refractory disease, second malignancy or death from any reason.

CONTACTS AND LOCATIONS:
Overall Officials: dunha zhou, M.D, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (9):
- China (9):
  - Maternal and Child Health Hospital of Foshan, Foshan, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangxi Province Children's Hospital Southern Medical University, China, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu LP, Zhang AL, Ruan M, Chang LX, Liu F, Chen X, Qi BQ, Zhang L, Zou Y, Chen YM, Chen XJ, Yang WY, Guo Y, Zhu XF. Prognostic stratification of molecularly and clinically distinct subgroup in children with acute monocytic leukemia. Cancer Med. 2020 Jun;9(11):3647-3655. doi: 10.1002/cam4.3023. Epub 2020 Mar 26. PMID 32216042
- [Result] Weis TM, Marini BL, Bixby DL, Perissinotti AJ. Clinical considerations for the use of FLT3 inhibitors in acute myeloid leukemia. Crit Rev Oncol Hematol. 2019 Sep;141:125-138. doi: 10.1016/j.critrevonc.2019.06.011. Epub 2019 Jun 28. PMID 31279288
- [Result] Rubnitz JE, Crews KR, Pounds S, Yang S, Campana D, Gandhi VV, Raimondi SC, Downing JR, Razzouk BI, Pui CH, Ribeiro RC. Combination of cladribine and cytarabine is effective for childhood acute myeloid leukemia: results of the St Jude AML97 trial. Leukemia. 2009 Aug;23(8):1410-6. doi: 10.1038/leu.2009.30. Epub 2009 Feb 26. PMID 19242495